CLINICAL TRIAL: NCT05967858
Title: Refeeding Syndrome - Incidence and Risk Factors: An Observational Study on Patients With G-I Disease and Head-neck Cancer
Brief Title: Incidence of Refeeding Syndrome in Consecutively Admitted Patients
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Assoc Prof, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: norge refeed
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Refeeding Syndrome; Starvation; Phosphate Deficiency
MeSH Terms: conditions — Refeeding Syndrome; Starvation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- gastroenterological: Consecutive admissions - n= 43 - 34 operated (79%) - 10 patients acutely admitted Diseases in Esophagus (8), gastric cavity (8), pancreas (7), colon/rectum (8), bile (4), small intestine (3), IBD (5) No interventions in the treatments, just observation
  Interventions: Other: observation
- head and neck cancer: Consecutive admissions - n=8 - 7 radiation therapy - 1 operated Locations: 2 Larynx, 1 oro-pharynx, 4 tonsillar, 1 tung No interventions in the treatments, just observation
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — no intervention

SUMMARY:
The incidence and main risk-factors analyzed in consecutive in-patients in the departments og gastroenterology and ear-nose and throat diseases (cancer in radiation therapy)

DETAILED DESCRIPTION:
Patients with either parenteral- or tube feeding enter the study to assure sufficient nutrition.

During hospitalization patients were monitored with daily blood samples and clinical evaluation of symptoms in addition to the coverage of energy and protein in percent of estimated needs.

Refeeding phenomenon was defined as a decrease in plasma phosphate after the initiation of nutrition.

Refeeding syndrome as refeeding phenomenon and one or more relevant symptoms in addition (hypotension, cardiac arrhythmia, edema, confusion)

ELIGIBILITY:
Inclusion Criteria:

* planned tube- or parenteral nutrition (complete or supplementary)
* > 18 years
* written consent

Exclusion Criteria:

* Renal insufficiency (p-creatinine >200 micromol/l)
* Lack of ability to communicate (registration of nutritional intake etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No other than willingness to participate and consecutively admitted, as well as planned sufficient nutrition
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Refeeding syndrome | 1 week after start of nutrition
  No. patients with decrease in plasma phosphate + clinical symptoms

SECONDARY OUTCOMES:
Refeeding phenomenon | 1 week after start of nutrition
  No. patients with decrease in plasma phosphate after start of nutrition

CONTACTS AND LOCATIONS:
Overall Officials: jens R Andersen, MD, MPA, Study Chair — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No